CLINICAL TRIAL: NCT05330494
Title: Effects of Perioperative Transcutaneous Electrical Acupoint Stimulation on Postoperative Pain and Agitation in Pediatric Adenoidectomy and Tonsillectomy
Brief Title: Effects of Perioperative TEAS on Postoperative Pain and Agitation in Pediatric Adenoidectomy and Tonsillectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xian Children's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2021-016-01
Record Dates: First submitted 2022-01-16; First posted 2022-04-15 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-05

CONDITIONS: the Effect of TEAS on the Children' Pain and Agitation
Keywords: Transcutaneous acupoint electrical stimulation; adenoidectomy; tonsillectomy; pain; agitation
MeSH Terms: conditions — Psychomotor Agitation; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- S1 (Experimental): TEAS treatment initiated at 30 minutes before induction and lasted for 30min,TEAS treatment(disperse-dense waves; frequency, 2/100 Hz)on acupoints Hegu(LI4) , Neiguan(PC6) and Zusanli（ST 36）of both sides, and the present intensity(8～12 mA) was the maximum current that could be tolerated.Then, the TEAS treatment was administered twice a day (once in the morning and once in the afternoon) on the first and second postoperative day, which lasted for 30 minutes each time.
  Interventions: Other: transcutaneous electrical acupoint stimulation(TEAS)
- S2 (Experimental): TEAS treatment initiated immediately after induction and stopped at the end of surgery,TEAS treatment(disperse-dense waves; frequency, 2/100 Hz)on acupoints Hegu(LI4) , Neiguan(PC6) and Zusanli（ST 36）of both sides, and the present intensity(8～12 mA) was the maximum current that could be tolerated.Then, the TEAS treatment was administered twice a day (once in the morning and once in the afternoon) on the first and second postoperative day, which lasted for 30 minutes each time.
  Interventions: Other: transcutaneous electrical acupoint stimulation(TEAS)
- S3 (Experimental): TEAS treatment initiated immediately after extubating and lasted for 30 minutes,TEAS treatment(disperse-dense waves; frequency, 2/100 Hz)on acupoints Hegu(LI4) , Neiguan(PC6) and Zusanli（ST 36）of both sides, and the present intensity(8～12 mA) was the maximum current that could be tolerated.Then, the TEAS treatment was administered twice a day (once in the morning and once in the afternoon) on the first and second postoperative day, which lasted for 30 minutes each time.
  Interventions: Other: transcutaneous electrical acupoint stimulation(TEAS)
- control (Sham Comparator): the control group was given all manipulations without electrical stimulation, electrodes were placed on the same acupoints, but no current was given
  Interventions: Other: transcutaneous electrical acupoint stimulation(TEAS)

INTERVENTIONS:
Other: transcutaneous electrical acupoint stimulation(TEAS) — transcutaneous electrical acupoint stimulation (TEAS), the modern therapies derived from traditional acupuncture, which could activate nerve endings or fibers and generate action potentials.s. TEAS uses self-adhesive electrodes placed on the surface of acupoints, instead of needles for electrical stimulation.The resulting stimulation signals, which are transmitted to the spinal cord and brain, stimulate the central nervous system to generate specific chemical mediators to induce relevant physiological effects.

SUMMARY:
Adenoidectomy and tonsillectomy are generally performed during childhood to help reduce snoring and improve sleep or caused by recurrent infection.And insufficient analgesia may result in postoperative sore throat, difficulty swallowing, aspiration, delayed discharge, spasm, and agitation. Remedial analgesic drugs such as morphine and opioids may lead to postoperative respiration depression, desaturation and vomiting.Transcutaneous electrical acupoint stimulation (TEAS) is a peripheral stimulation, which is a modern therapy derived from traditional acupuncture. Relevant clinical trials show that it can effectively relieve pain, and has slight side-effects.However, most of these clinical trials are conducted in adults, and there have been few clinical trials involving children. For this reason, in line with good tolerance and less side effects of TEAS, ,this study is designed to enhance the therapeutic effect of adenoidectomy and tonsillectomy pain by means of taking advantage of the skin-sticking electro-acupuncture.It is also hoped that this study can certify if TEAS can reduce the amount and side effects of analgesic drugs, such as morphine, and improve the postoperative safety of children, and moreover, explore the possible mechanisms by which TEAS relieve pain in children.

DETAILED DESCRIPTION:
Sample size The sample size estimation was based on the incidence of agitation in previous studies. It was selected for a type I error of 0.05, a power of 0.80, and the dropout rate 0f 0.2. The calculation was done through a website program (https://www.medsci.cn), and 200 patients should be included .

Randomization and blinding On arrival at the operating room, a simple randomization method will be used to make sure that the patient is randomly allocated to one of four groups at the 1:1:1:1 ratio.Investigator put the group information in four different envelopes. When the first envelope is extracted, the following patients intelligently extract the group from the remaining envelopes, and so on, until all four envelopes are extracted, and investigator repeat the process. The anesthesiologist who carried out the TEAS procedures and in charge of intraoperative anesthesia is aware of the assignment to group TEAS. But the outcome assessors responsible for collecting and analyzing the data are blind to patient treatment.

Procedure Before entering the operating room, intravenous (IV) access should be clear and no medication is given previously. After entering the operating room, electrocardiogram (ECG), pulse oxygen inundation (SpO2), noninvasive blood pressure (NIBP), SedLine and analgesia nociception index(ANI) are checked according to the manufacturer's recommendations . At the same time, the electrodes are placed at Hegu (LI4), Neiguan （PC 6）and Zusanli (ST36) of both sides.Anesthesia is induced with 2-3 mg/kg of propofol, 0.3 µg/kg of sufentanil. Meanwhile, 0.1 mg/kg of atropine and 0.2 mg/kg of dexamethasone are given to prevent postoperative nausea and oral secretions. After confirming the absence of a response to eye stimulus, 0.15 mg/kg of cis-atracurium is administered. Ventilation is conducted with a mask using 100% oxygen, and tracheal intubation is done after realizing the adequate depth of anesthesia. Next, to preserve the spectral edge frequency (SEF) between 14 and 20, anesthesia is maintained with the end-tidal concentration of sevoflurane 2-2.5 vol% and remifentanil at a dose of 0.2-0.3ug/kg/min during surgery, while ventilation is measured to sustain the end-tidal carbon dioxide (EtCO2) between 40 ± 5 mmHg. Furthermore, baseline hemodynamic variations are kept within a ±20% range.

Intervention patients are randomly divided into TEAS and control groups, and TEAS group is divided into three subgroups (S1, S2 and S3) according to the time of treatment started: S1 treatment initiate at 30 minutes before induction and last for 30min, S2 treatment initiate immediately after induction and stop at the end of surgery, S3 treatment initiate immediately after extubating and last for 30 minutes. The TEAS group receive TEAS treatment(disperse-dense waves; frequency, 2/100 Hz)on acupoints Hegu(LI4) , Neiguan(PC6) and Zusanli（ST 36）of both sides, and the present intensity(8～12 mA) is the maximum current that could be tolerated. Then, the TEAS treatment is administered twice a day (once in the morning and once in the afternoon) on the first and second postoperative day, which last for 30 minutes each time. And the control group is given all manipulations without electrical stimulation.

Statistical analyses Measurement data of normal distribution are reported as the mean ± SD. Categorical variables are analyzed through chi-squared test or the Fisher's exact probability test and presented as numbers (%). Comparisons between two groups are performed with Student's t-test. Repeated measurements were compared using repeated measure' ANOVA. For all tests, P<0.05 is considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. the American Society of Anesthesiologists physical status Ⅰ and Ⅱ.
2. Ranging in age from 4 to 10.
3. Suffering from adenoid and/or tonsil hypertrophy
4. Preparing for elective surgery under general anesthesia with a signed written informed consent by parents..

Exclusion Criteria:

1. immunological, neurological, and hematological disorders
2. having any drug allergy or asthma, as well as allergic constitution
3. with congenital heart disease or various malignant arrhythmias
4. skin infections existing at acupoints and their surroundings
5. history of receiving acupuncture or electroacupuncture treatment
6. long-term use of analgesic or sedative drugs
7. used to having unilateral tonsil ablation
8. refusing to join the trial investigator
9. postoperative trachea spasm or laryngeal edema occurring

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2022-04-25 (Actual); Primary Completion 2022-10-30 (Estimated); Study Completion 2023-03-10 (Estimated)

PRIMARY OUTCOMES:
change from pain score within 48 hours after surgery | interval 5minutes for the first 30 minutes after extubation, and then for the outstanding 24 hours and 48 hours after surgery
  it is caused by procedure , and assessed with the Face, Legs, Activity, Cry, Consolability （FLACC ）pain scale,a higher score indicates more severe pain
change from agitation score within 48 hours after surgery | interval 5 minutes for the first 30 minutes after extubation, and then for the outstanding 24 hours and 48 hours after surgery
  postoperative agitation is a reformed state of mindfulness, which starts with a sudden form of anesthesia and progresses through the early repossession age,it is assessed with the Pediatric Anesthesia Emergence Delirium (PAED) scale.It includes five objects (eye contact with the caregiver, purposeful action, and awareness of surroundings, restlessness, and inconsolability). Each item was scored by five scores (0 to 4) permitting to its degree, for a maximum of 20 points.Agitation was defined as a PAED 10 points.

SECONDARY OUTCOMES:
duration of anesthesia | Intraoperative (from the start of induction to endotracheal tube (EET) removal)
  the time required for anesthesia from induction to completion
duration of surgery | Intraoperative (from the insertion of the mouth gag to removal of the mouth gag)
  the time required for an operation from start to finish
recovery time | Intraoperative (from sevoflurane discontinuation to spontaneous eye opening)
  the time it takes to wake up from sevoflurane discontinuation
extubation time | Intraoperative (from discontinuation of sevoflurane to tracheal extubation)
  the time from discontinuation of sevoflurane to tracheal extubation, and endotracheal tube was uninvolved when breathing was steady and adequate in rate and depth
PACU length of stay(PACU-LOS) | up to 48 hours (from the time patients' arrival in PACU to the time leaving PACU after surgery)
  patient's stay time in PACU
postoperative length of stay(PLOS) | from the date of operation to the date of discharge , an average of 3 days
  The time between the date of operation and discharge in the hospital
the concentration of serum interleukin-6 (IL-6), cortisol (COR) and β-endorphin(β-EP) | entering the operating room, 30minutes after extubation, 24 hours after surgery
  blood samples were extracted to detect the concentration of serum interleukin-6 (IL-6), cortisol (COR) and β-endorphin(β-EP) at the time of entering the operating room, 30minutes after extubation, 24hours after surgery
change from mean arterial pressure (MAP) on the day of surgery | Intraoperative (entering the operating room, just before induction, intubation, insertion of the mouth gag, removal of the mouth gag, 0 minute, 5 minutes, 10 minutes, 15 minutes, 30 minutes after extubation)
  refers to the noninvasive mean arterial pressure,the average of arterial blood pressure over a cardiac cycle
change from heart rate (HR) on the day of surgery | entering the operating room, just before induction, intubation, insertion of the mouth gag, removal of the mouth gag, 0 minute, 5 minutes, 10 minutes, 15 minutes, 30 minutes after extubation
  number of heart beats per minute
change from analgesia nociception index(ANI) on the day of surgery | entering the operating room, just before induction, intubation, insertion of the mouth gag, removal of the mouth gag, 0 minute, 5 minutes, 10 minutes, 15 minutes, 30 minutes after extubation
  derived from heart rate variability,it is a proposed guide to obtain an adequate control of the analgesic component during anaesthesia,the higher the pain index, the worse the pain relief
the consumption of remifentanil | Intraoperative (From the beginning to the end of the operation)
  remifentanil dosage during the procedure
postoperative sufentanil rescue rate in PACU | up to 48 hours (from the time patients' arrival in PACU to the time leaving PACU after surgery)
  sufentanil was given at a dose of 0.1ug/kg when the patient's pain score was greater than or equal to 4 in PACU
the incidence of postoperative nausea and vomiting(PONV) | from the end of surgery to 48 hours after surgery
  The incidence of postoperative nausea and vomiting in four groups
postoperative sleep quality | 24hours and 48 hours after surgery
  Postoperative sleep status of patients,it is assessed with the Pittsburgh Sleep Quality Index (PSQI) questionnaire，0~5 good sleep quality，6~10 sleep quality is ok,11 to 15 average sleep quality,16 to 21 poor sleep quality
complications | from end of surgery to 48 hours after operation
  various adverse events occurred after operation

CONTACTS AND LOCATIONS:
Overall Officials: Fang Li Yang, Study Chair — Xi 'an children's hospital
Locations (1):
- Xi'an Children's Hospital, Xi'an, Shaanxi, China